CLINICAL TRIAL: NCT05871580
Title: Effect to the Photobiomodulation in the Burning Mouth Syndrome. A Randomised Doble-Blind Clinical Trial.
Brief Title: Effect to the Photobiomodulation in the Burning Mouth Syndrome
Acronym: PBM-BMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT-PBM/BMS-23
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Burning Mouth Syndrome; Quality of Life; Anxiety Depression; Dry Mouth
Keywords: Burning Mouth Syndrome; Oral Manifestations; Quality of Life; Anxiety Depression; Hyposalivation; Xerostomia
MeSH Terms: conditions — Burning Mouth Syndrome; Xerostomia; Oral Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: One group will be lasered off and the other group will be lasered on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (GL) (Active Comparator): The patients will be submitted to eight sessions of low power laser. The radiation emission will be performed according to the protocol.
  Interventions: Radiation: Low frequency laser activated photobiomodulation
- Control Group (CG) (Placebo Comparator): In these patients the investigators will use the same protocol applied in the experimental group (time and application values) but the laser device will be turn off.
  Interventions: Other: Low frequency laser photobiomodulation inactive

INTERVENTIONS:
Radiation: Low frequency laser activated photobiomodulation — Infravermelho: analgesia, tissue biostimulation. The number of laser application points will be determined based on the areas referred by the patients.
  * apex tongue: 3 points
  * lateral edge of the tongue: 4 points
  * tongue dorsum: 10 points
  * jugal mucosa: 8 points
  * labial mucosa: 5 points
  * hard palate: 8 stitches
  * soft palate: 3 stitches
  * gingiva or alveolar mucosa: 3 stitches per sextant.
  Time of 30 seconds in each application point, with dosage: 3 J/point.
  Arms: Laser Group (GL)
Other: Low frequency laser photobiomodulation inactive — The same protocol as the activated group
  Arms: Control Group (CG)

SUMMARY:
Introduction: Burning mouth syndrome (BMS) is a pathology with a low prevalence, affecting between 0.1% and 3.7% of the general population, the ratio between women and men is between 3 and 7:1. It is clinically characterized by a burning pain sensation, recurrent daily for more than 2 hours a day, persistent for more than 3 months and in a way that increases throughout the day and decreases at night, without presenting clinically evident causal lesions on the surface of the oral mucosa, nor changes in clinical sensory tests.

The description of the symptomatology varies according to the patient and may be related especially to psychogenic factors.

Patients report dry mouth/xerostomia and taste alterations, such as metallic or bitter taste. The most frequent location is on the tongue (tip and lateral borders), but it can also include the anterior palate, gingiva and lips.

Since the etiopathogenic factors that produce BMS are not clear, it is difficult to make advances in therapy. The available treatments aim to control the multiple factors related to BMS, thus reducing the symptoms described by patients. Among them, the literature describes low level laser photobiomodulation.

The success of the use of low level lasers for treatments in oral medicine is due to their biomodulatory activity and their ability to penetrate tissues. The analgesic action of laser radiation is due to the inhibition of nociceptive mediators and the release by the Central Nervous System (CNS) of endogenous analgesic substances such as endorphins, which hinders the transmission of the painful stimulus.

It has been verified that low power laser radiation therapy can be effective in reducing symptoms in patients with BMS. Importantly, low power laser therapy is non-invasive, well tolerated by patients.

Objectives: To confirm the hypothesis that the application of low power laser in the areas of oral burning can improve the symptomatology of BMS.

Material and methods: We propose a clinical study in 38 patients with idiopathic BMS, prospective, randomized, double-blind.

The study universe will be constituted by patients attended at the Oral Medicine, Oral Surgery and Implantology Unit of the Faculty of Dentistry of the University of Santiago de Compostela (USC).

The Hospital Anxiety and Depression Scale (HADS), quality of life (OHIP-14) and subjective sensation of dry mouth xerostomia inventory (XI) questionnaires will be applied to all the patients, and the amount of saliva will be quantitatively determined by means of the unstimulated global saliva test (TSG-I) using a millimetric absorbent paper strip, at the beginning, at the end of treatment and at the re-evaluation at two and six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of BMS and symptoms of at least 3 months duration;
* Clinical examination confirms clinically normal mucosa;
* Patients who are not undergoing treatment for BMS;
* Patients who, after being informed about the objectives and procedures of the investigation, agree and sign the informed consent form.

Exclusion Criteria:

* Patients with uncontrolled systemic diseases (ASA III, IV);
* Patients who have received previous radio and/or chemotherapy of the head and neck;
* Patients with secondary BMS, which is due to organic causes, such as biological factors, i.e. the presence of some bacteria or fungi, which have a direct irritant effect on the oral mucosa and are capable of triggering burning symptoms. Such conditions considered as differential diagnosis of primary BMS which are, oral candidiasis, erosive lichen planus, geographic tongue;
* Patients presenting systemic factors such as Sjögren's syndrome, untreated diabetes, or if they use drugs that cause oral burning;
* Patients presenting a VAS score below 3 out of 10.

Removal criteria:

-Patients who for any reason fail to keep follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Pain reported | 6 months
  To evaluate the effect of 808 nm diode laser radiation (infrared) applied intraorally on areas where patients report burning mouth. The degree of pain/burning reported by patients using a visual analogue scale (VAS). Scale from 0 to 10, where zero means no pain and ten means severe pain.

SECONDARY OUTCOMES:
Degree of anxiety of the patients | 6 months
  To evaluate the degree of anxiety of the patients, through the Hospital Anxiety and Depression Scale (HADS). For every question the patient must answer about the presence or frequency of the symptoms, with four possible answers. The score ranges from 0 to 3 points for every question, depending on the intensity of the symptoms. Therefore, the total HADS score ranges from 0 to 21 points for each subscale.
Quality of life of the patients | 6 months
  Assess quality of life, using OHIP-14. For scoring the answers to each of the 14 questions in the OHIP-14, the following values are used: 0 = never, 1 = rarely, 2 = sometimes, 3 = frequently, 4 = always, with the maximum possible score reaching 56 points.
Subjective sensation of dry mouth | 6 months
  Assess the subjective sensation of dry mouth through the xerostomia inventory.
Quantitative measurement of saliva | 6 months
  Quantitative measurement of saliva through the unstimulated global saliva test (TSG-I).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group.